CLINICAL TRIAL: NCT01462565
Title: A Single-arm, Open Label Study Evaluating the Impact on Lifestyle of a New Thermo Stable Formulation of FLOLAN® in Subjects With Pulmonary Arterial Hypertension (PAH). (FLOLAN® is a Registered Trademark of the GlaxoSmithKline Group of Companies.)
Brief Title: Study of a New Thermo Stable Formulation of Epoprostenol Sodium to Treat Pulmonary Arterial Hypertension (PAH)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115332
Record Dates: First submitted 2011-10-13; First posted 2011-10-31 (Estimated); Results first posted 2017-10-16 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-05

CONDITIONS: Hypertension, Pulmonary
Keywords: flolan; pulmonary arterial hypertension; thermo stable formulation; epoprostenol sodium; modified sterile diluent
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — Epoprostenol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All subjects (Experimental): Subjects enter the study already taking current marketed FLOLAN (epoprostenol sodium) and continue for 4 weeks (run-in). At baseline, they will be swopped to the new thermo stable formulation of epoprostenol sodium for 4 weeks (or longer if they continue in the extension phase of the study).
  Interventions: Drug: current marketed FLOLAN (epoprostenol sodium); Drug: new thermo stable formulation of epoprostenol sodium

INTERVENTIONS:
Drug: current marketed FLOLAN (epoprostenol sodium) — continuous intravenous infusion
Drug: new thermo stable formulation of epoprostenol sodium — continuous intravenous infusion

SUMMARY:
The purpose of this multicentre, open label, single-arm study in approximately 20 adult patients is to evaluate the Impact on lifestyle of a new thermo stable formulation of epoprostenol sodium in subjects with Pulmonary Arterial Hypertension (PAH).

DETAILED DESCRIPTION:
This is a multicentre, open label, single-arm study in approximately 20 adult patients (18 - 75 years old) designed to evaluate the Impact on lifestyle of a new thermo stable formulation of epoprostenol sodium in subjects with Pulmonary Arterial Hypertension (PAH). The co-primary objectives are 1) to describe the effect of the new thermo stable formulation of epoprostenol sodium on quality of life and 2) to determine the dose titration requirement in patients switching from the currently marketed FLOLAN (epoprostenol sodium) to the new thermo stable formulation. Secondary objectives include assessing the safety, tolerability and efficacy of the thermo stable formulation of epoprostenol sodium and the exploratory objective is to evaluate the effect of the new thermo stable formulation of epoprostenol sodium on haemodynamic parameters in a subset of subjects.

Subjects who are already receiving FLOLAN (epoprostenol sodium) for the treatment of PAH and have been on a stable dose for at least 3 months and on stable doses of other PAH treatments for at least 30 days prior to screening will be enrolled. After a screening visit, eligible subjects will have a 4-week run-in period with their existing FLOLAN (epoprostenol sodium) treatment. At the end of the 4-week period, they will be admitted to the clinic for baseline assessments and for switching to study medication (the new thermo stable formulation of epoprostenol sodium). Subjects will remain in hospital for a minimum of 6 hours to ensure clinical and hemodynamic stability prior to discharge. Subjects may stay in hospital for up to 24-48 hours after switching to the new thermo stable formulation of epoprostenol sodium at the discretion of the investigator. Dose titration requirement will be assessed at the time of discharge. Haemodynamic parameters will be obtained in a subgroup of subjects enrolled in centres where the collection of haemodynamic data is considered part of the standard of care. Subjects will receive the study medication as a continuous intravenous infusion for a 4-week treatment period. Those who complete the 4-week treatment period will have the option of entering an extension phase of the study to continue receiving the new formulation.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female at least 18 to 75 years at the time of screening.
* Subjects must have been on FLOLAN (epoprostenol sodium) therapy for pulmonary arterial hypertension (PAH) as approved in the product label.
* Subjects must be on stable doses of their existing FLOLAN (epoprostenol sodium) treatment for a minimum of 3 months prior to screening.
* Subjects must be on stable doses of any current PAH treatments other than FLOLAN (epoprostenol sodium) in the last 30 days.
* Subjects must walk a distance of at least 150 meters during six-minute walk distance test (6MWD). This test must be completed during the Screening Visit.
* A female subject is eligible to participate if she is of non-childbearing potential or of childbearing potential, has a negative pregnancy test at screen, and agrees to use one of the contraception methods listed in the protocol.
* Subjects must be competent to understand the information given in the Institutional Review Board (IRB) or Independent Ethics Committee (IEC) approved informed consent form and must sign the form prior to the initiation of any study procedures.

Exclusion Criteria:

* Subjects who are given FLOLAN (epoprostenol sodium) for a condition or in a manner that is outside the approved indication.
* Subjects with congestive heart failure arising from severe left ventricular dysfunction.
* Subjects, with or without supplemental oxygen, who have a resting arterial oxygen saturation (SaO2) <90% as measured by pulse oximetry at screening.
* Subjects have been hospitalized as an emergency or visited the emergency room for a condition related to PAH or treatment for PAH in the last 3 months.
* The subject's clinical condition is such that they are not expected to remain clinically stable for the duration of the study.
* Female subjects who are pregnant or breastfeeding.
* Subjects who have demonstrated noncompliance with previous medical regimens.
* Subjects who have a history of abusing alcohol or illicit drugs within 1 year.
* Subjects with a diagnosis of active hepatitis (hepatitis B surface antibody and hepatitis C antibody).
* Subjects who have participated in a clinical study involving another investigational drug or device within four weeks before screening.
* Subjects who had history malignancies within the past 5 years, with the exception of basal cell carcinoma of the skin or in situ carcinoma of the cervix.
* Any concurrent condition that would affect the safety of the subject or in the opinion of the investigator it is not in the best interest of the patient to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-11-01; Primary Completion 2012-05-16 (Actual); Study Completion 2012-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- United States (6):
  - GSK Investigational Site, Miami Beach, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Dallas, Texas
- GSK Investigational Site, Québec, Quebec, Canada
- GSK Investigational Site, Amsterdam, Netherlands

REFERENCES:
- [Derived] Provencher S, Paruchuru P, Spezzi A, Waterhouse B, Gomberg-Maitland M; pH12 Flolan reformulation study group. Quality of life, safety and efficacy profile of thermostable flolan in pulmonary arterial hypertension. PLoS One. 2015 Mar 20;10(3):e0120657. doi: 10.1371/journal.pone.0120657. eCollection 2015. PMID 25793960

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 17 participants were recruited from 23 November 2011 to 16 May 2012, out of which 16 participants entered the treatment phase. Study was conducted across 5 centres in the United States, 1 centre in Canada and 1 centre in the Netherlands.
Pre-assignment Details: There was a 4-week run-in period during which 1 participant was assessed to be a screen failure at the Baseline Visit (Visit 2) due to the participant self-titrating their epoprostenol sodium. During the 4-week run-in period, participants received currently marketed epoprostenol sodium.
Groups:
- Epoprostenol Sodium for Injection: Participants received new thermo stable 100 milliliter (mL) formulation of epoprostenol sodium via intravenous infusion each day for 4-week treatment period.
Period: Overall Study
Arm/Group | Epoprostenol Sodium for Injection
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Epoprostenol Sodium for Injection: Participants received new thermo stable 100 mL formulation of epoprostenol sodium via intravenous infusion each day for 4-week treatment period.
Arm/Group | Epoprostenol Sodium for Injection
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.0 (13.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Medical Outcomes Study Short Form 36 (SF-36)
Description: Subject-rated measure of health status comprised of 36 items: 8 subscale scores (physical functioning, role limitations due to physical health problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health), 2 summary scores (physical component and mental component), and a self-evaluated change in health status. Subscale and summary scores range: 0-100. Higher subscale and summary scores was considered as better health status. Change from Baseline was calculated as score at observation minus score at baseline. Baseline was defined as Visit 2 i.e. Day-14 (+ or - 7 days).
Time Frame: Baseline (Visit 2 i.e. Day-14 [+ or - 7 days]) and Week 4 (Visit 3)
Population: Intent-to-Treat (ITT) population consisted of all participants who received at least one dose of epoprostenol sodium during the Run-in period (either currently marketed epoprostenol sodium or the study drug).
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Epoprostenol Sodium for Injection
Number analyzed (Participants) | 16
Score on a scale
  Physical Functioning | -1.156 (3.6593)
  Role-Physical | -0.765 (6.3050)
  Role-Emotional | 0.002 (11.1773)
  Vitality | 0.781 (7.1636)
  Mental Health | 0.883 (7.6063)
  Social Functioning | 1.706 (7.1043)
  Bodily Pain | 3.065 (5.8291)
  General Health | -0.606 (5.6068)
  Physical Health Component | -0.123 (4.2876)
  Mental Health Component | 1.141 (6.5078)

2. Primary Outcome: Change From Baseline in Study Specific Participant Acceptance Survey
Description: Study-specific questionnaire comprised the pre-defined15 questions which included activities of daily living assessment. Participants rated the question on a scale of 1 to 10, where 1 was do not agree and 10 was strongly agree. Change from Baseline was calculated as score at observation minus score at Baseline. Changes from Baseline was assessed for Questions 2 to 12. Baseline was defined as Visit 2 i.e. Day-14 (+ or - 7 days).
Time Frame: Baseline (Visit 2 i.e. Day-14 [+ or - 7 days]) and Week 4 (Visit 3).
Population: ITT population.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Epoprostenol Sodium for Injection
Number analyzed (Participants) | 16
Score on a scale
  Q2- ability to perform physical activities | -0.9 (2.29)
  Q3- ability to perform your basic daily activies | -1.5 (1.86)
  Q4- ability to perform activities with your family | -0.8 (2.37)
  Q5- ability to participate in social activities | -0.9 (1.88)
  Q6- ability to comply with your Flolan treatment | 0.3 (3.34)
  Q7- ability to perform new activity(Jogging, walk) | 0.4 (2.00)
  Q8- overall satisfaction | 0.4 (1.09)
  Q9- interested physical activity | -0.1 (2.53)
  Q10- feel physically restricted from participating | 0.1 (2.73)
  Q11- confident in my ability to do new activity | 0.6 (2.50)
  Q12- treatment regimen constantly weighs on mind | -0.6 (1.75)

3. Primary Outcome: Change From Baseline in Dose of Thermo Stable Epoprostenol Sodium at Week 4
Description: Dose titration requirement was assessed at the time of discharge. Change from Baseline was calculated as score at observation minus score at Baseline. Units- nanogram per kilogram per minute (ng/kg/min). Baseline was Visit 2 i.e . Day-14 (+ or - 7 days).
Time Frame: Baseline (Visit 2 i.e. Day-14 [+ or - 7 days]) and Week 4
Population: ITT population.
Measure: Mean (Standard Deviation); unit: ng/kg/min
Arm/Group | Epoprostenol Sodium for Injection
Number analyzed (Participants) | 16
ng/kg/min | 0.22 (1.169)

4. Secondary Outcome: Number of Participants With Any Treatment Emergent Adverse Events (AEs) and Treatment Emergent Serious Adverse Events(SAEs)
Description: An AE was defined as any untoward medical occurrence that occurred during the course of the trial after study treatment had started. An adverse event was therefore any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. An SAE is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, congenital anomaly/birth defect and medically significant and all events of possible drug-induced liver injury with hyperbilirubinaemia. Only treatment emergent AEs and SAEs were reported in this outcome measure. Specifically, this study reported 2 SAEs, but only 1 was categorized as treatment emergent.
Time Frame: Up to visit 3 (Week 4)
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoprostenol Sodium for Injection
Number analyzed (Participants) | 16
Participants
  Any AEs | 9
  Any SAEs | 1

5. Secondary Outcome: Number of Participants With Infusion Site Reactions During Treatment Period
Description: Infusion site reactions were reported during the treatment period. Infusion site was inspected for erythema, excoriation, induration, skin necrosis or signs of local sepsis.
Time Frame: Baseline visit (Visit 2) to Week 4 (Visit 3)
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoprostenol Sodium for Injection
Number analyzed (Participants) | 16
Participants
  Erythema | 1
  Signs of local sepsis | 1
  Other | 1

6. Secondary Outcome: Change From Baseline in Vital Signs at Week 4 : Systolic and Diastolic Blood Pressure
Description: Systolic blood pressure is a measure of blood pressure while the heart is beating. Diastolic blood pressure is a measure of blood pressure while the heart is relaxed. Change from Baseline was calculated as the value at the indicated time points minus the value at Baseline. Baseline was Visit 2 i.e. Day-14 (+ or - 7 days).
Time Frame: Baseline (Visit 2 i.e. Day-14 [+ or - 7 days]) and Week 4(Visit 3)
Population: ITT population.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Epoprostenol Sodium for Injection
Number analyzed (Participants) | 16
Millimeter of mercury (mmHg)
  Systolic blood pressure | -0.4 (11.47)
  Diastolic blood pressure | 0.4 (10.99)

7. Secondary Outcome: Change From Baseline in Vital Signs at Week 4: Heart Rate
Description: Summary mean change in heart rate measured in beats per minute (beats/min or BPM). Change from Baseline was calculated as the value at the indicated time points minus the value at Baseline. Baseline was Visit 2 i.e. Day-14 (+ or - 7 days).
Time Frame: Baseline (Visit 2 i.e. Day-14 [+ or - 7 days]) to Week 4
Population: ITT population.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Epoprostenol Sodium for Injection
Number analyzed (Participants) | 16
beats/min | -1.7 (8.52)

8. Secondary Outcome: Number of Participants With Abnormal Clinical Chemistry
Description: Abnormal clinical chemistry was analyzed as follows: serum alanine aminotransferase (ALT/SGPT) >= 3 x upper limit of normal (ULN) , aspartate aminotransferase (AST/SGOT) >= 3 x ULN , total bilirubin >= 34.2, creatinine >= 176.8.
Time Frame: Up to 1 week after Week 4 (Follow-up)
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoprostenol Sodium for Injection
Number analyzed (Participants) | 16
Participants | 0

9. Secondary Outcome: Number of Participants With Abnormal Hematology
Description: Values for hemoglobin, hematocrit, and platelet count were analyzed. Participants with abnormal values have been reported. The low and high value concern were as follows: hemoglobin (Males < 98, >180.0) (females <91, >161.0)grams per litre (g/L); hematocrit (Males < 32.0, >54.0) (females <29.0, >50.6) fraction (1); platelet count (< 100, > 500) gram international units per litre (gI/L).
Time Frame: Up to 1 week after Week 4 (Follow-up)
Population: ITT population. Only those participant available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoprostenol Sodium for Injection
Number analyzed (Participants) | 16
Participants
  Hemoglobin (G/L) : Week 4: high: number analyzed (Participants) | 15
  Hemoglobin (G/L) : Week 4: high | 1
  Hematocrit (1): Screening: Low: number analyzed (Participants) | 14
  Hematocrit (1): Screening: Low | 14
  Hematocrit (1): Baseline: Low: number analyzed (Participants) | 15
  Hematocrit (1): Baseline: Low | 15
  Hematocrit (1): Week 4: Low: number analyzed (Participants) | 15
  Hematocrit (1): Week 4: Low | 15
  Hematocrit (1): Follow-up: Low: number analyzed (Participants) | 1
  Hematocrit (1): Follow-up: Low | 1
  Platelet count (GI/L): Screening: Low: number analyzed (Participants) | 14
  Platelet count (GI/L): Screening: Low | 5
  Platelet count (GI/L): Baseline: Low: number analyzed (Participants) | 13
  Platelet count (GI/L): Baseline: Low | 2
  Platelet count (GI/L): Week 4: Low: number analyzed (Participants) | 14
  Platelet count (GI/L): Week 4: Low | 1
  Platelet count (GI/L): Follow up: Low: number analyzed (Participants) | 1
  Platelet count (GI/L): Follow up: Low | 1

10. Secondary Outcome: Number of Participants With Abnormal Urinalysis
Description: Dipstick method was used to measure blood, glucose and protein. Data was analyzed up to 1 week after Week 4 (Follow-up visit).
Time Frame: Up to 1 week after Week 4 (Follow-up)
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoprostenol Sodium for Injection
Number analyzed (Participants) | 16
Participants | 0

11. Secondary Outcome: Change From Baseline in Six Minute Walk Distance Test (6MWD) After 4-weeks of Treatment
Description: This assessment was a non-encouraged test that measures the distance walked for a duration of 6 minutes. Change from Baseline was calculated as value at observation minus value at Baseline. Baseline visit was Visit 2 i.e. Day-14 (+ or - 7 days).
Time Frame: Baseline (Visit 2 i.e. Day-14 [+ or - 7 days]) and Week 4
Population: ITT population.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Epoprostenol Sodium for Injection
Number analyzed (Participants) | 16
meters | -3.55 (45.321)

12. Secondary Outcome: Breathlessness After 6MWD - Borg Dyspnoea Index (BDI)
Description: The BDI was calculated by using a 10-point scale (0 = None, 10 = Maximum) and indicates the degree of breathlessness after completion of the 6-minute walk test. The BDI scale was assessed by each participant. Change from Baseline = score at observation minus score at Baseline. Baseline visit was Visit 2 i.e. Day-14 (+ or - 7 days).
Time Frame: Baseline (Visit 2 i.e. Day-14 [+ or - 7 days]) to Week 4
Population: ITT population.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Epoprostenol Sodium for Injection
Number analyzed (Participants) | 16
Score on a scale | 0.36 (0.535)

13. Secondary Outcome: World Health Organization [WHO] Functional Class at Baseline and After 4- Weeks of Treatment
Description: World Health Organization functional class was analyzed as class I, class II, class III and class IV. World Health Organization functional class was analyzed at Baseline (Visit 2 i.e. Day-14 [+ or - 7 days]) and Week 4. The classed were defined as Class I: No symptoms of pulmonary arterial hypertension with exercise or at rest, Class II: No symptoms at rest but uncomfortable and short of breath with normal activity, Class III: May not have symptoms at rest but activities greatly limited by shortness of breath, fatigue, or near fainting and Class IV: Symptoms at rest and severe symptoms with any activity. Hence the severity increased from class I (better) to Class IV (worse).
Time Frame: Baseline (Visit 2 i.e. Day-14 [+ or - 7 days]) and Week 4
Population: ITT population. Only those participants with data available at the specified time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoprostenol Sodium for Injection
Number analyzed (Participants) | 16
Participants
  Baseline WHO Class I: number analyzed (Participants) | 15
  Baseline WHO Class I | 2
  Baseline WHO Class II: number analyzed (Participants) | 15
  Baseline WHO Class II | 9
  Baseline WHO Class III: number analyzed (Participants) | 15
  Baseline WHO Class III | 4
  Baseline WHO Class IV: number analyzed (Participants) | 15
  Baseline WHO Class IV | 0
  Week 4 Class I | 2
  Week 4 Class II | 10
  Week 4 Class III | 4
  Week 4 Class IV | 0

14. Secondary Outcome: Mean Oxygen Saturation in Blood Over Time
Description: Pulse oximetry (oxygen saturation) was analyzed. Data for Pulse oximetry (oxygen saturation) was analyzed up to the treatment follow up (1 week after Visit 3 [Week 4]).
Time Frame: up to the treatment follow up (1 week after Visit 3 [Week 4])
Population: ITT population. Only those participant available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of oxygen in blood
Arm/Group | Epoprostenol Sodium for Injection
Number analyzed (Participants) | 16
Percentage of oxygen in blood
  Baseline | 94.3 (1.95)
  Week 4 | 94.5 (2.58)
  Follow-up (1 week after Week 4): number analyzed (Participants) | 1
  Follow-up (1 week after Week 4) | 93.0 (NA) — Data for only 1 participant was analyzed.

15. Secondary Outcome: Number of Participants With Urine Pregnancy Test Positive
Description: Urine samples were collected for urine pregnancy test. Urine samples were collected at up to the treatment follow up (1 week after Visit 3 [Week 4]). Number of participants with urine pregnancy test positive has been reported.
Time Frame: up to the treatment follow up (1 week after Visit 3 [Week 4])
Population: ITT population. Only those participants with data available at the indicated time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoprostenol Sodium for Injection
Number analyzed (Participants) | 12
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to 1 week after Week 4 (Follow-up) for SAEs and Up to Visit 3 (Week 4) for non-serious adverse events.
Description: ITT population was used for the analysis of AEs and SAEs.
Arm/Group | Epoprostenol Sodium for Injection
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 2/16
Other Adverse Events (participants affected / at risk) | 9/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Epoprostenol Sodium for Injection (N=16)
Device related infection (Infections and infestations) | 2
Catheter site haemorrhage (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Epoprostenol Sodium for Injection (N=16)
Ascites (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Paraesthesia oral (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Oedema peripheral (General disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Bronchitis (Infections and infestations) | 1
Catheter site infection (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Headache (Nervous system disorders) | 2
Thyroiditis (Endocrine disorders) | 1
Haematoma (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.